CLINICAL TRIAL: NCT04491500
Title: Retinal and Choroidal Circulation Changes Following Rapid Ascent to a High Altitude Environment Evaluated by OCT Angiography
Brief Title: Retinal and Choroidal Circulation Changes Following Rapid Ascent to a High Altitude Environment
Status: Completed | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shanshan Yu, MD, Clinical Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2020051
Record Dates: First submitted 2020-07-22; First posted 2020-07-29 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: High Altitude Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: This is a self-control study. Subjects who plan togo to 4000m altitude to work for two weeks will be enrolled. And before and after they arrive high altitude, they will have visual acuity, OCTA, and intraocular pressure; blood pressure, blood oxygen measurement.
  Interventions: Behavioral: High attitude environment

INTERVENTIONS:
Behavioral: High attitude environment — The participants will go to 4000m altitude to work for two weeks.

SUMMARY:
This is a prospective observational study. The purpose is to explore the effect of high altitude hypobaric hypoxia on retinal microcirculation and the change of the thickness of the retina and choroid by optical coherence tomography angiography (OCTA).

DETAILED DESCRIPTION:
Yushu is in Qinghai-Tibet plateau, an average altitude of 4000 m. The medical staff is limited in Yushu. Zhongshan ophthalmic center, sun yat-sen university in Yushu blindness project has lasted many years. Some medical staff who arrived at Yushu will have a plateau response. The high altitude hypoxia on retinal microcirculation evaluated by OCTA has not been reported. The aim of the study is to observe the microcirculation changes after exploring a hypobaric and hypoxia environment using OCTA, and relation with the plateau response. OCTA is a non-invasive examination and could see the microcirculation of the fundus directly and quickly.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects who plan to go to Yushu within one month.
2. Did not live on the high altitude of more than 1000 meters within 6 months.

Exclusion Criteria:

1. Unable and unwilling to provide informed consent.
2. Any ocular disease may influence the retinal and choroidal circulation.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: the staff will go to Yushu on the 2020 preventive blindness project.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
retinal microcirculation changes | 1 month
  the vascular density measured by OCTA

SECONDARY OUTCOMES:
Retinal thickness changes | 1 month
  the retinal thickness measured by OCTA
Choroidal thickness changes | 1 month
  the subfoveal choroidal thickness measured by OCTA
The correlation of retinal microcirculation with the altitude illness | 1 month
  The relationship between retinal vascular density as measured by OCTA and the degree of altitude illness as measured by acute mountain sickness (AMS) scoring system
The changes of intraocular pressure | 1 month
  The changes of intraocular pressure measured by icare Tonometer
The changes of blood pressure including systolic and diastolic Blood Pressure | 1 month
  The changes of blood pressure measured by Blood Pressure Meter
The changes of blood oxygen | 1 month
  The changes of blood Oxygen measured by Pulse Oximeter
the degree of altitude illness | 1 month
  the degree of altitude illness was assessed by acute mountain sickness (AMS) scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Liang, M.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Liang xiaoling, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
After the result publish online, the data will be shared.